CLINICAL TRIAL: NCT01084993
Title: EArly Discharge After Transradial Stenting of CoronarY Arteries in High-Risk Patients of Bleeding: Bivalirudin to Reduce Bleeding EASY-B2B Study
Brief Title: EArly Discharge After Transradial Stenting of CoronarY Arteries in High-Risk Patients of Bleeding
Acronym: EASY-B2B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Olivier F. Bertrand, MD, PhD, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EASY-B2B
Record Dates: First submitted 2010-03-09; First posted 2010-03-11 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery stenting, transradial, intracoronary
MeSH Terms: conditions — Coronary Artery Disease | interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bivalirudin (Active Comparator): Standard practice: 0.75mg/kg + infusion 1.75mg/kg/h
  Interventions: Drug: Bivalirudin
- Heparin (Active Comparator): 70 U/kg or standard practice
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin — Standard practice: 0.75mg/kg + infusion 1.75mg/kg/h
  Other Names: Angiomax
  Arms: Bivalirudin
Drug: Heparin — 70 U/kg
  Arms: Heparin

SUMMARY:
RATIONALE:

Transradial coronary stenting is associated with less risk of access site complications and bleeding compared to femoral approach.

Major bleeding post-PCI is a strong independent predictor of mortality and MACE. Depending of the antithrombotic regimen and access-site used, bleeding related to access-site represents 50-80% of the cases. Whereas transradial approach minimizes the risks of access-site bleeding, it has no impact on non-access site bleeding.

Peri-procedural anemia is also an independent predictor of mortality and MACE.

With femoral approach, bivalirudin compared to heparin ± glycoproteins IIb-IIIa has been associated with a significant reduction in access-site and non-access site related bleeding.

In a post-hoc analysis of patients treated by transradial approach in ACUITY, there was a trend for non-access site bleeding (organ bleeding) with bivalirudin compared to heparin ± glycoproteins IIb-IIIa.

HYPOTHESES:

In patients at high-risk of peri-procedural bleeding, bivalirudin ± glycoproteins IIb-IIIa reduces the risk of bleeding compared to heparin ± glycoproteins IIb-IIIa.

In patients at high-risk of bleeding and undergoing transradial PCI, bivalirudin significantly reduces the incidence of non-access site bleeding and peri-procedural anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary objective is to compare the incidence of major bleeding and anemia 24h post-PCI in patients at high-risk of bleeding after transradial PCI with heparin or bivalirudin.

ELIGIBILITY:
Inclusion Criteria:

* At least two of the following additional criteria
* At least 70 yrs old
* Female gender
* Diabetes
* Creatinine clearance <60mL/min
* History of gastro-intestinal or other organ bleeding
* Baseline anemia
* Current treatment with glycoproteins IIb-IIIa inhibitors

Exclusion Criteria:

* Intolerance or allergy to ASA, clopidogrel or ticlopidine precluding treatment for 12 months
* Concurrent participation in other investigational study
* Femoral sheath (artery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2010-03; Primary Completion 2018-09 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Major bleeding and Mace | 24h post-PCI and Discharge
  The primary end-points will be 1) the incidence of major bleeding (Replace-2 criteria) at hospital discharge and 2) the incidence of 24h post-PCI anemia (WHO criteria)

SECONDARY OUTCOMES:
EFFICACY and SAFETY PARAMETERS | 30 days
  The composite of death, MI (def 1 : Tn-t > 0.1 and def 2 : CK-MB > 30μg/l), urgent revascularization and major bleeding at 30 days post-PCI.
  The incidence of ARC-defined stent thrombosis at 30 days. The incidence of access-site hematoma according to EASY scale. The incidence of radial artery occlusion at hospital discharge according to echo-doppler evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD, PhD, Principal Investigator — Fondation IUCPQ
Locations (1):
- Quebec Heart-Lung Institute, Québec, Quebec, Canada